CLINICAL TRIAL: NCT05879185
Title: Phase II Study of XmAb23104 (Targeting PD-1 and ICOS), in Patients With Advanced Sarcoma
Brief Title: A Study of XmAb23104 in People With Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Vendor decided study to be closed early
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-195
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sarcoma
Keywords: XmAb23104; PD-1; ICOS; 22-195
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: This phase II, open-label, single-center study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XmAb23104 in People With Sarcoma (Experimental): Patients will receive the recommended phase II dose of XmAb23104 monotherapy on day 1 and 15 of each 28-day cycle. Patients will continue XmAb23104 (day 1 & 15, q 28 days) for up to 24 months depending on their response and tolerability to treatment. Treatment will be continued until progressive disease (PD) or toxicity or a total of 24 months of study therapy has been completed.
  Interventions: Biological: XmAb23104

INTERVENTIONS:
Biological: XmAb23104 — XmAb23104 (10 mg/kg) intravenously on days 1 and 15 of each 28-day cycle. XmAb23104 will be administered by IV infusion at a constant rate over 1 hour.

SUMMARY:
The purpose of this study is to find out whether the study drug, XmAb23104, is an effective treatment for advanced sarcoma. The researchers will also look at whether XmAb23104 is safe and causes few or mild side effects in participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years at the time of informed consent
* Be capable, willing, and able to provide written informed consent/assent
* Be willing to comply with clinical trial instructions and requirements, including mandatory biopsies at baseline and on-treatment where feasible
* Patients must have progressed on or be intolerant of at least one prior standard systemic therapy where available. If a patient declines standard systemic therapy they will be considered eligible.
* Patients must have a histologically confirmed locally advanced/metastatic sarcoma with select histological subtypes including

  * i) malignant solitary fibrous tumor (SFT)
  * ii) leiomyosarcoma (LMS)
  * iii) dedifferentiated chondrosarcoma
  * iv) undifferentiated pleomorphic sarcoa/myxofibrosarcoma (Patients with UPS/MFS will be eligible if they have refractory to or relapsed after anti-PD-(L)1 therapy and demonstrated clinical benefit to immunecheckpoint inhibition [complete/partial response or stable disease >/=6 months])
  * v) sclerosing epithelioid fibrosarcoma (SEF) or extraskeletal myxoid chondrosarcoma (ESMC)
  * vi) pecoma.
* Adequate performance status: ECOG 0 or 1/KPS 100-70%
* Expected life expectancy >3 months
* Presence of measurable disease per RECIST v1.1.

  o Target lesion(s) must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment
* Adequate organ function determined within 10 days of treatment initiation

  * Platelet count > 100 x 10^9/L
  * Hemoglobin level > 8.0 g/dL
  * Absolute neutrophil count > 1.0 x 10^9/L
  * AST at screening < 3 x ULN for subjects without known liver involvement by tumor; or < 5 x ULN for subjects with known liver involvement by tumor
  * ALT at screening < 3 x ULN for subjects without known liver involvement by tumor; or < 5 x ULN for subjects with known liver involvement by tumor
  * Bilirubin ≤ 1.5 × ULN (unless prior diagnosis and documentation of ongoing hemolysis or Gilbert's syndrome has been made)
  * Estimated creatinine clearance (CL) > 30 mL/min calculated by the Cockcroft-Gault or modification of diet in renal disease formulas
* Female subjects of childbearing potential must agree to use a highly effective method of birth control during and for 8 weeks after completion of study. Women are considered to be of childbearing potential unless it is documented that they are over the age of 60 OR postmenopausal by history with no menses for 1 year and confirmed by FSH OR have a history of hysterectomy and/or bilateral oophorectomy OR have a history of bilateral tubal ligation. Highly effective methods of birth control include hormonal birth control (oral, intravaginal, transdermal, implantable, or intrauterine device [IUD]), IUDs (non-hormonal), vasectomy (in male partner), or any double-barrier methods (combination of male condom and spermicide with either cap, diaphragm, or sponge).

Exclusion Criteria:

* History of unstable or deteriorating cardiovascular disease within the previous 6 months prior to screening including but not limited to the following:

  * Unstable angina or myocardial infarction
  * CVA/stroke
  * Congestive heart failure (New York Heart Association [NYHA] Class III or IV
  * Uncontrolled clinically significant arrhythmias
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Patients with previously treated brain metastases or carcinomatous meningitis may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases on imaging performed during study screening, and are not using steroids for at least 14 days prior to trial treatment
* Current use of immunosuppressive medication, EXCEPT for the following:

  * intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 2 months prior to enrollment
* History or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 years prior to enrollment. Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease
* A life threatening (Grade 4) immune related adverse event related to prior immunotherapy.
* Failure to recover from any immune related adverse event from prior anti-cancer therapy to grade ≤ 1, with the exception of alopecia or endocrinopathies that are managed and stable on hormone replacement therapy.
* Failure to recover from any other toxicity (other than immune-related toxicity) related to previous anticancer treatment to Grade ≤ 2 except for alopecia and peripheral neuropathy related to prior chemotherapy
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) disease that is not controlled HIV positive patients will be considered eligible if:

  * Established ART for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment
  * CD4+ T-cell (CD4+) counts ≥ 350 cells/uL
  * No opportunistic infection within the past 12 months
* Patients known to be positive for active Hepatitis B (HBsAg reactive with detectable HBV DNA), or Hepatitis C (HCV RNA (qualitative) is detected)

  * Patients with chronic hepatitis B (positive HBsAg and/or HBcAb and negative HBV DNA by PCR) are eligible for this study if they are on suppressive anti-viral therapy and deemed safe by a gastroenterologist
  * Patient who is HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution will be considered eligible.
* Has a known history of active TB (Bacillus Tuberculosis)
* Women who are pregnant or breastfeeding
* Patients expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment(s)
* Prior organ transplantation including allogenic stem-cell transplantation
* Active infection requiring systemic therapy
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5 Grade ≥ 3)
* Prior treatment with an investigational anti-ICOS therapy
* Treatment with a PD-1 or PD-L1 antibody within 8 weeks of the start of study therapy.
* Treatment with any other anticancer therapy within 3 weeks of the start of study drug (ie, other immunotherapy, chemotherapy, radiation therapy, etc.).
* Treatment with antibiotics within 14 days prior to first dose of study drug
* Receipt of a live-virus vaccine within 30 days prior to first dose of study drug (vaccines that do not contain live virus are permitted).
* Presence of any other active malignancy requiring systemic therapy that may influence the outcome of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
best objective response rate | 24 weeks
  by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ciara Kelly, MBBCh BAO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm